CLINICAL TRIAL: NCT04304755
Title: Zoledronic Acid as Adjuvant Therapy in Neovascular Age-related Macular Degeneration (The Z-AMD Study): A Randomized Controlled Pilot Study
Brief Title: Zoledronic Acid as Adjuvant Therapy in Neovascular Age-related Macular Degeneration (Z-AMD)
Acronym: Z-AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Morten Carstens Moe, MD, Professor in Ophthalmology, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/583
Record Dates: First submitted 2020-02-23; First posted 2020-03-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: zoledronic acid; anti-VEGF; anti-vascular endothelial growth factor; adjuvant therapy; AMD
MeSH Terms: interventions — Zoledronic Acid; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Medical Product : Zoledronic acid (Experimental): Zoledronic acid 5 mg IV at baseline and after 26 weeks.
  Interventions: Drug: Zoledronic Acid 5 MG in 5 ML Injection
- Placebo: NaCl 0,9% (Placebo Comparator): 100 ml 0.9% NaCl IV at baseline and after 26 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Zoledronic Acid 5 MG in 5 ML Injection — Zoledronic acid
  Other Names: ZA
  Arms: Investigational Medical Product : Zoledronic acid
Drug: Placebos — NaCl 0.9%
  Other Names: NaCl
  Arms: Placebo: NaCl 0,9%

SUMMARY:
A pilot study of zoledronic acid as adjuvant therapy to standard anti-vascular endothelial growth factor (anti-VEGF) treatment for neovascular age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This is a one-year, randomized, controlled pilot study. A total of 40 treatment-naïve nAMD patients will be allocated 1:1 to receive an intravenous infusion of either zoledronic acid (ZA) 5 mg or placebo at baseline and after 26 weeks as adjuvant therapy to intravitreal anti-VEGF injections in accordance with a treat and extend algorithm; bevacizumab is the first-line treatment, and refractory eyes are converted to aflibercept.

The participants will be recruited among patients admitted to the Department of Ophthalmology at Oslo University Hospital (OUH). The department is the largest provider of retinal care in Norway and serves a local community of almost one million people, which makes it well-suited for recruitment. Administration of ZA or placebo will take place at Pilestredet Park Specialist Centre, an endocrinology clinic in Oslo with particular interest in treatment of osteoporosis. The Clinical Trial Unit at OUH will monitor the study.

ELIGIBILITY:
Inclusion Criteria:

1. Active, treatment-naïve neovascular AMD in the study eye, intraretinal or subretinal fluid involving the fovea centre on optical coherence tomography (OCT), and evidence of choroidal neovascularization on fluorescein angiography (FA) and/or OCT angiography (OCT-A).
2. Age ≥50 years
3. Best-corrected visual acuity (BCVA) between 0.1 and 1.0 logMAR
4. Menopausal for at least one year
5. Only one eye per patient will be recruited for the study. If both eyes are eligible for the study, the eye with the wors best-corrected Visual acuity (BCVA) will be selected as the study eye.
6. Subjects must give written informed consent before any study related procedures are performed

Exclusion Criteria:

1. Lesions comprising more than 50% blood or fibrosis involving the fovea centre
2. Polypoidal choroidal vasculopathy (PCV) - indocyanine green (ICG) angiography is performed at the discretion of the investigator on clinical suspicion of PCV
3. Presence of other ocular disease causing concurrent vision loss
4. Presence of ocular disease making intravitreal treatment contraindicated (e.g. current ocular or periocular infection, active uveitis or uncontrolled glaucoma/intraocular pressure ≥ 25 mmHg)
5. Systemic anti-vascular endothelial growth factor (anti-VEGF) or bisphosphonate treatment within one year preceding the initial study treatment
6. Confirmed or suspected active malignancy
7. Other factors (i.e. lack of cooperation) that, in the opinion of the investigator, can interfere with the study protocol
8. Known or suspected hypersensitivity to any of the trial products
9. Hypocalcemia (total Ca < 2.15 mmol/L)
10. Renal impairment (estimated ClCR < 35 ml/min).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in best-corrected visual acuity (BCVA) after 52 weeks. | 52 weeks
  To assess the change in best-corrected visual acuity measured by logMAR.

SECONDARY OUTCOMES:
The number of anti-VEGF intravitreal injections given after 52 weeks | 52 weeks
  To assess the number of anti-VEGF injections needed during 52 weeks of treatment.
Number of patients with a change in BCVA of 0.3 logMAR or more after 52 weeks. | 52 weeks
  Number of patients with a change in BCVA of 0.3 logMAR or more after 52 weeks.
Proportion of patients with refractory nAMD after 52 weeks. | 52 weeks
  Proportion of patients with refractory nAMD after 52 weeks.
EQ 5D score (ranging from 0-1; 0 designates "perfect health" and NEI-VFQ-25 score (ranging from 0 to 100 where 100 reflects best vision-specific health). | 52 weeks
  EQ 5D score (ranging from 0-1; 0 designates "perfect health" and NEI-VFQ-25 score (ranging from 0 to 100 where 100 reflects best vision-specific health).
Mean change from baseline in Central retinal thickness (CRT) after 52 weeks. | 52 weeks
  Mean change from baseline in Central retinal thickness (CRT) after 52 weeks.To assess the proportion of patients with a considerable change in visual function
Proportion of patients experiencing adverse events of special interest (ESI): osteonecrosis of the jaw or atypical femoral fracture, endophthalmitis or orbital, scleral, or serious intraocular inflammation (grade 4 aqueous cells/FLARE). | 52 weeks
  Proportion of patients experiencing adverse events of special interest (ESI): osteonecrosis of the jaw or atypical femoral fracture, endophthalmitis or orbital, scleral, or serious intraocular inflammation (grade 4 aqueous cells/FLARE).

CONTACTS AND LOCATIONS:
Overall Officials: Morten C Moe, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Spesialistsenteret Pilestredet Park, Oslo
  - Oslo university hospital, Department of Ophthamology, Oslo

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04304755/SAP_000.pdf